CLINICAL TRIAL: NCT04994964
Title: Pilot Study of Recurrent Laryngeal Nerve Monitoring During Neonatal Aortic Arch Repair
Brief Title: Recurrent Nerve Monitoring During Aortic Arch Repair
Acronym: PREMAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 20/BC/CARDIO/NO/444
Record Dates: First submitted 2021-03-11; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-04

CONDITIONS: Recurrent Laryngeal Nerve Injuries; Aortic Arch Hypoplasia
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries | interventions — Electromyography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electromyography — Needle vocal cord electromyography using Medtronic NIM monitor

SUMMARY:
Almost half of newborns undergoing surgery to repair narrowing or interruption of the aortic arch will suffer injury to the recurrent laryngeal nerve. This causes a weak voice and can lead to problems with feeding including aspiration of milk feed after the surgery. As these children can have a vulnerable circulation, aspiration events can reduce survival and poor weight gain has been shown to correlate with poorer outcomes after surgery.

In other types of surgery in the neck, monitors can be used to alert the surgeon to when injury is occurring to the recurrent nerve. To date, this type of monitoring has not been possible in newborns. This study aims to investigate if this type of monitoring is feasible in newborns undergoing aortic arch repair, to prevent recurrent nerve injury.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with parents/ carers able to give informed consent to participation in the trial will be included. • Male and female patients will be included
* Only Neonates (babies less than 28 days of age) will be included in the study.
* Only patients undergoing repair of the aortic arch via median sternotomy will be included in the study

Exclusion Criteria:

* Patients with severe abnormalities of the airway, such that they are unlikely to be extubated within 7 days of the aortic arch repair surgery will be excluded from participation, as assessment of vocal cord function will be difficult/ impossible in such patients.
* Patients with parents/ carers who are unable to give informed consent to participation in the trial will be excluded from participation.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Vocal cord EMG - Burst amplitude (mV) | Intra-operative (1 hour)
  Feasibility of performing vocal cord EMG during neonatal arch repair
Vocal cord EMG - Burst duration (ms) | Intra-operative (1 hour)
  Feasibility of performing vocal cord EMG during neonatal arch repair
Vocal cord EMG - Burst frequency (Hz) | Intra-operative (1 hour)
  Feasibility of performing vocal cord EMG during neonatal arch repair
Vocal cord EMG - Interburst interval (ms) | Intra-operative (1 hour)
  Feasibility of performing vocal cord EMG during neonatal arch repair
Vocal cord EMG - Signal to noise ratio (mV) | Intra-operative (1 hour)
  Feasibility of performing vocal cord EMG during neonatal arch repair
Correlation of Vocal cord EMG with post-operative palsy | Post extubation / 1 week post-operatively
  Vocal cord ultrasound

SECONDARY OUTCOMES:
Neuromuscular blockade | Intra-operative (1 hour)
  Influence of timing of neuromuscular blockade on EMG signal

CONTACTS AND LOCATIONS:
Overall Officials: Phil Botha, PhD, Principal Investigator — Birmingham Women's and Children's Hospital
Locations (1):
- Birmingham Children's Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No